CLINICAL TRIAL: NCT03412968
Title: Using Polysulfone Membranes on Continuous Ultrafiltration With Volume Replacement in Patients Undergoing Cardiac
Brief Title: Continuous Hemofiltration During Cardiopulmonary Bypass and Its Effect on Lactatemia
Acronym: CPB-LACTATE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Cadiz (Other)
Collaborators: Mª José Abellán Hervás (Unknown); Rocío Martín Valero (Unknown); Ana María Sáinz Otero (Unknown)
Responsible Party: Principal Investigator, Carlos Garcia Camacho, MSc, University of Cadiz
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 160/16
Record Dates: First submitted 2018-01-16; First posted 2018-01-29 (Actual); Last update posted 2018-05-11 (Actual); Status verified 2018-05

CONDITIONS: Cardiovascular Diseases
MeSH Terms: conditions — Cardiovascular Diseases | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Intervention Model Description: The perfusionist's role is essential during the procedure involving Cardiopulmonary Bypass (CPB). This study purpose to know the impact of using polysulfone membranes on continuous ultrafiltration with volume replacement in patients undergoing cardiac surgery. In this type of surgery, techniques such as conventional ultrafiltration (CUF) and modified ultrafiltration (MUF) are known for controlling the patient's fluid balance and blood lactate levels during the procedure.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Polysulfone Filter Group (Experimental): The purpose of the research is to determine whether, by controlling the patient's hemodilution level and, therefore, the acute anaemia caused by the Cardiopulmonary Bypass (CPB) priming fluid, continuous conventional ultrafiltration (CUF) can decrease serum lactate levels during normothermic CPB by increasing the haematocrit and, consequently, the supply of oxygen to the tissues, and whether the haemofiltration membrane can remove lactate molecules in situations of hyperlactataemia in CPB.
  Interventions: Procedure: Polysulfone Filter
- Control Group (Active Comparator): The purpose of the research is to determine serum lactate levels during normothermic cardiopulmonary bypass procedure (CPB) without continuous hemofiltration of the patient during the CPB.
  Interventions: Procedure: Procedure/ Surgery: without Polysulfone Filter

INTERVENTIONS:
Procedure: Polysulfone Filter — The intervention for this group consisted using a Polysulfone filter in order to hemofiltration in the procedure involving Cardiopulmonary Bypass (CPB).The perfusionist's role is essential during the procedure, as they control both Cardiac Output (CO) and gas exchange, depending on their action, will affect blood lactate levels.
  Arms: Polysulfone Filter Group
Procedure: Procedure/ Surgery: without Polysulfone Filter — In this group, no intervention is performed during the procedure involving Cardiopulmonary Bypass (CPB)
  Arms: Control Group

SUMMARY:
This study aims to analyze the impact of using polysulfone membranes on continuous ultrafiltration with volume replacement in patients undergoing cardiac surgery. In this type of surgery, techniques such as conventional ultrafiltration (CUF) and modified ultrafiltration (MUF) are known for controlling the patient's fluid balance during the procedure. However, there is no scientific evidence on the benefits of continuous haemofiltration with volume replacement and its effect on lactatemia. Method and design: A single center randomized controlled trial, parallel treatment design with patient-blinded to compare outcomes in terms of the lactate clearance rates (quantity/unit of time) of the assigned therapy groups. Participants will be randomly assigned to receive the type of surgery, in order to ensure an unbiased assessment of treatments, randomisation will be performed in eight blocks of five patients. The study groups will be equivalent in all aspects except the procedures they undergo. Participants will be assigned to the first control group without haemofiltration (CG or 1) or one group with haemofiltration using a Polysulfone filter (PG or 2). Data will be collected by a blinded evaluator.

DETAILED DESCRIPTION:
To determine whether continuous ultrafiltration with volume replacement using a polysulfone membrane during Cardiopulmonary Bypass (CPB) in patients undergoing cardiac surgery decreases intraoperative lactatemia.

ELIGIBILITY:
Inclusion Criteria:

* Patients who signed informed consent
* Patients not undergoing emergency surgery.
* Surgical procedures performed under normothermic conditions.
* Patients with a minimum time of 40 minutes before decannulation (after the end of myocardial reperfusion, unclamping of the aorta and the end of CPB).

Exclusion Criteria:

* Emergency medical condition in which it is not possible to collect study data.
* Heart condition requiring the use of hypothermia or hyperthermia during CPB.
* Patients without a minimum time of 40 minutes before decannulation (after the end of myocardial reperfusion, unclamping of the aorta and the end of CPB).
* Patients who cannot manage their fluid balance on their own through diuresis prior to CPB.
* Patients who are unable to manage excess volume during the surgical procedure by means of spontaneous or forced diuresis with diuretics (positive cumulative balance despite intravenous bolus of diuretics after 75% of the anticipated duration of CPB according to the course of the surgery).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2018-01-30 (Actual); Study Completion 2018-02-28 (Actual)

PRIMARY OUTCOMES:
Plasma Lactate Level | Baseline
  The lactate level will be measured before Cardiopulmonary Bypass (CPB) in all patients

SECONDARY OUTCOMES:
Maximum Plasma Lactate Level | Every 20 minutes from the start of the Cardiopulmonary Bypass (CPB)
  The maximum level of intraoperative lactate will be measured in all patients, whether the polysulfone membrane has been used or not during Cardiopulmonary Bypass (CPB)
Plasma Lactate Level | 1 minute after the Cardiopulmonary Bypass (CPB)
  The level of lactate level will be measured in all patients, whether the polysulfone membrane has been used or not at the end cardiopulmonary bypass (CPB).
Plasma Lactate Level in the effluent | 1 minute after the Cardiopulmonary Bypass (CPB)
  To determine lactate levels in the effluent in all ultrafiltered patients
Plasma Lactate Level in intensive care unit (ICU) | 24 hours after the Cardiopulmonary Bypass (CPB)
  Lactate level will be measured 24 hours after surgery in ICU stay
Serum potassium Level | Every 20 minutes from the start of the Cardiopulmonary Bypass (CPB)
  Serum potassium level measured in routine analysis blood
Evaluation criteria of mortality and risk profiles of population | 10 minutes before the Cardiopulmonary Bypass (CPB)
  Mortality predicted and operative risk will be measured by scoring systems European System for Cardiac Operative Risk Evaluation (EuroSCORE I) in cardiac surgery in all patients
Hematocrit | Every 20 minutes from the start of the Cardiopulmonary Bypass (CPB)
  Hematocrit measured in routine analysis blood in all patients

CONTACTS AND LOCATIONS:
Overall Officials: Carlos García Camacho, Degree, Principal Investigator — University of Cadiz; María José Abellán Hervás, PhD, Study Director — University of Cadiz; Rocío Martín Valero, PhD, Study Director — University of Cadiz; Ana María Sáinz Otero, Study Director — University of Cadiz
Locations (1):
- Hospital Puerta del Mar, Cadiz, Spain